CLINICAL TRIAL: NCT03193008
Title: Current Value of Axillary Ultrasound in the Staging of Breast Cancer. Is BSGC Still Necessary?
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Javier del Riego, MD, Corporacion Parc Tauli
Other Study IDs: CPT-JDR-2017-1
Record Dates: First submitted 2017-04-28; First posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Axillary ultrasound; Sentinel lymph node biopsy; Axillary management
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
AUS/FNAC allows the identification of tumors without axillary tumor involvement, or with low axillary tumor burden, many of which do not benefit from SLNB, in the staging of early breast cancer.

Objective: To calculate the negative predictive value of AUS/FNAC in those patients with breast cancer who meet ACOSOG Z0011 criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Tumors with ACOSOG Z0011 criteria, except positive SLNB (cT1-T2; cN0; breast-conserving surgery; Whole-Breast Radiotherapy)
* Axillary study with AUS/FNAC.
* SLNB/ALND (Gold-Standard).

Exclusion Criteria:

* Tumors without confirmation of axillary histologic status (No Gold-Standard)
* Tumor in pregnancy or breastfeeding.
* Tumors in the male.
* Tumors treated with neoadjuvant chemotherapy
* Tumors that do not meet ACOSOG Z0011 criteria.
* Tumors without axillary study using AUS/FNAC

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed breast cancer from January 2008 to December 2013
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-07-15 (Estimated); Study Completion 2017-07-15 (Estimated)

PRIMARY OUTCOMES:
Detection of axillary tumor burden by axillary ultrasound | Two weeks after the axillary surgery
  To calculate the negative predictive value of AUS/FNAC in those patients with breast cancer who meet ACOSOG Z0011 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Javier del Riego, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No